CLINICAL TRIAL: NCT07259122
Title: A Phase II Clinical Study of Zanubrutinib Combined With Four Cycles of CD20 Monoclonal Antibody and Reduced-Dose Bendamustine in the Treatment of Untreated Waldenström Macroglobulinemia
Acronym: ZBR in WM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025111
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Waldenström Macroglobulinemia (WM)
Keywords: zanubrutinib; bendamustine
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bendamustine Hydrochloride; Rituximab; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: ZBR (Experimental)
  Interventions: Drug: Zaunbrutinib, Bendamustine and Rituximab for induction therapy; Drug: Zanubrutinib mono therapy for maintenance treatment

INTERVENTIONS:
Drug: Zaunbrutinib, Bendamustine and Rituximab for induction therapy — Patients in the experimental group will receive treatment in 4-week cycles, totaling 4 cycles of zanubrutinib + bendamustine + CD20 Monoclonal Antibody therapy, followed by 8 months of zanubrutinib monotherapy maintenance.
  Specific regimen:
  Zanubrutinib: Oral administration starts on Day 1 of Cycle 1 and continues continuously at 160 mg twice daily.
  Bendamustine: Intravenous infusion at 70 mg/m² on Days 1-2 of Cycles 1-4. CD20 Monoclonal Antibody: Intravenous infusion at 375 mg/m² on Day 0 of Cycles 1-4.
  After completing the 4-cycle combination therapy, a systematic efficacy evaluation will be conducted.
Drug: Zanubrutinib mono therapy for maintenance treatment — Patients will then continue with zanubrutinib monotherapy maintenance for 8 months before treatment discontinuation.

SUMMARY:
This study is a prospective phase II clinical trial designed to evaluate the deep response rate of the ZBR regimen (zanubrutinib combined with reduced-dose bendamustine and CD20 Monoclonal Antibody ) in treatment-naïve symptomatic Waldenström macroglobulinemia (WM) patients. Eligible patients will receive four cycles of the ZBR regimen, followed by zanubrutinib monotherapy for an additional eight months. The assessment period spans from the initiation of treatment until 12 months after treatment completion, with efficacy evaluations conducted every three cycles. Patients will be withdrawn from the study if they experience disease progression (PD) or show no response to treatment. Minimal residual disease (MRD) assessments will be performed at the end of the 3rd and 6th treatment cycles, as well as 12 months after treatment completion, involving evaluations of both bone marrow and peripheral blood MRD rates

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female patients aged ≥18 years.
* 2. Must meet the diagnostic criteria for Waldenström's Macroglobulinemia (WM).
* 3. Patients must be treatment-naïve or not have received standard prior therapy, as defined by the following conditions: a) No prior combined chemotherapy with regimens such as BR, RCD, BCD, CHOP, or COP. b) No prior therapy with fludarabine-containing regimens. c) Treatment with chlorambucil or cyclophosphamide (alone or in combination with glucocorticoids) for less than 4 weeks. d) Failure to achieve a minimal response (MR) from the above treatments. e) If any of the above treatments were previously administered, a washout period of at least 2 weeks must be completed before study treatment initiation.
* 4. Presence of indications for WM treatment, meeting at least one of the following criteria: a) Symptomatic hyperviscosity. b) Symptomatic peripheral neuropathy. c) Amyloidosis. d) Cold agglutinin disease; cryoglobulinemia. e) Disease-related cytopenia (Hemoglobin <100 g/L or Platelet count <100×10^9/L). f) Massive lymphadenopathy. g) Presence of constitutional symptoms: persistent/recurrent fever (>38°C) for over 2 weeks unrelated to infection, drenching night sweats, and/or unintentional weight loss >10% within 6 months. h) Rapid disease progression, defined as a >50% increase in lymph node size within 2 months, and/or lymphocyte doubling time <6 months, and/or rapid decline in hemoglobin or platelet counts not due to autoimmune causes. i) Evidence of histologic transformation.
* 5. ECOG Performance Status score of ≤2.
* 6. Laboratory values meeting the following criteria within the screening period: Absolute Neutrophil Count (ANC) ≥ 0.75 × 10^9/L; Platelet count ≥ 50 × 10^9/L; Total Bilirubin ≤ 2 × Upper Limit of Normal (ULN); Alanine Aminotransferase (ALT) / Aspartate Aminotransferase (AST) ≤ 3 × ULN; Calculated creatinine clearance ≥ 30 mL/min (using Cockcroft-Gault formula)
* 7. Life expectancy of ≥ 6 months.

Exclusion Criteria:

* 1. Diagnosis or treatment for any malignancy other than B-cell non-Hodgkin lymphoma (B-NHL) within the past year (including active central nervous system lymphoma).
* 2. Clinical evidence of transformation to large cell lymphoma.
* 3.Pre-existing severe hepatic or renal impairment unrelated to lymphoma: ALT > 3 × ULN; AST > 3 × ULN; Total Bilirubin > 2 × ULN; Estimated creatinine clearance < 30 mL/min
* 4.Any other severe concurrent medical condition that would, in the investigator's judgment, compromise the patient's ability to participate in the study (e.g., uncontrolled diabetes, gastric ulcer, significant cardiac or pulmonary disease, etc.). The final determination rests with the investigator.
* 5. Known history of human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) infection, or any uncontrolled active systemic infection requiring intravenous antibiotic therapy. Note: Active HBV infection is defined by ALL of the following criteria: a. HBV DNA ≥ 2000 IU/mL; b. ALT ≥ 2 × ULN; c. Hepatitis not attributable to other causes such as the underlying disease or drugs. Patients with initially active HBV who convert to an inactive carrier state after antiviral therapy may be enrolled if they receive adequate concomitant antiviral prophylaxis.
* 6. Symptomatic central nervous system dysfunction or involvement (Bing-Neel syndrome).
* 7. Major surgery within 14 days prior to the first dose of study drug or anticipated requirement for major surgery during the study treatment period (excluding lymph node biopsy).
* 8. Inability to swallow capsules, or conditions significantly affecting gastrointestinal function (e.g., malabsorption syndrome, status post-gastrectomy or small bowel resection, symptomatic inflammatory bowel disease, ulcerative colitis, partial or complete intestinal obstruction).
* 9. Requirement for concurrent strong Cytochrome P450 (CYP) 3A inhibitors.
* 10. Pregnancy or lactation. Women of childbearing potential unwilling to use effective contraception during the study period.
* 11. Known hypersensitivity to any of the study drugs or their excipients.

Withdrawal Criteria

* 1. Disease progression during treatment (after ≥2 cycles of therapy) or failure to achieve at least a minimal response (MR) after 6 cycles of therapy.
* 2. Occurrence of intolerable adverse events or complications.
* 3. Patient's voluntary decision to withdraw consent for continued treatment.
* 4. Pregnancy during the study.
* 5. Investigator's judgment that the patient should discontinue treatment for any other reason.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Best deep response rate(≥VGPR) | up to 1 year
  defined as the rate of very good partial response VGPR or CR

SECONDARY OUTCOMES:
MRD Negativity Rate at End of Treatment | up to the end of treatment
  MRD Negativity Rate at End of Treatment
Duration of Response | up to 3 years
  The length of time between the achievement of criteria for response to treatment (first documented complete or partial response) and the first documented relapse or progression.
Objective Response Rate (ORR) | up to 1 year
  Response Rate (ORR) is defined as the proportion of subjects who achieve CR ,VGPR, PR or MR at the end of Treatment
Complete Response (CR) Rate | up to 1 year
  To assess CR rate at the end of treatment
Major Response Rate (MRR, ≥ Partial Response) | up to 1 year
  Response Rate (ORR) is defined as the proportion of subjects who achieve CR or PR at the end of Treatment
Time to First Response | up to 1 year
  Time to First Observed Response During Treatment
Time to Best Response | up to the end of treatment
  Time to the Best Response
Progression-Free Survival (PFS) | up to 3 years
  The time from the enrollment of a subject to the occurrence of (in any way) progression of disease or Death for any reason. patients with indeterminate recurrence or Death at the last follow-up, defined as the date of the last Investigation
Overall Survival (OS) Rate | up to 3 years
  The time from subject enrollment to Death caused by any reason. for patients lost to follow-up, the time of the last follow-up; for patients still alive at the end of study, the date of the end of follow-up.
Time to Next Treatment (TTNT) | up to 3 years
  Time from the initiation of the current treatment regimen to the start of the next line of therapy
Treatment-Related Adverse Events (AEs) | up to 3 years
  Incidence of adverse events, serious adverse events and significant adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Yi, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (2):
- China (2):
  - China Institute of Hematology and Blood Diseases Hospital ,Chinese Academy of Medical Sciences, Tianjin, China
  - Institute of Hematology & Blood Diseases Hospital, China, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No